CLINICAL TRIAL: NCT04437108
Title: Efficacy of Low-intensity Shock Wave Therapy on Persistent Storage Symptoms After Transurethral Surgery for Benign Prostatic Obstruction: A Randomized Controlled Trial
Brief Title: Efficacy of Li-SWT on Persistent Storage Symptoms After Transurethral Surgery for BPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Ahmed Mohamed Elshal (Unknown)
Responsible Party: Principal Investigator, Mohammed Hegazy, assistant lecturer of urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Li-SWT after relief of BPO
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Overactive Bladder; Urinary Incontinence, Urge; Urgency-frequency Syndrome; Post Prostatectomy
Keywords: low-intensity shock wave therapy; persistent storage symptoms; benign prostatic obstruction
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Li-SWT (Active Comparator): Patients will be treated by 8 sessions of Li-SWT with one week interval. This group is subdivided into 3 subgroups according to the approach through which Li-SWT is applied; suprapubic, perineal and combined approaches
  Interventions: Procedure: Li-SWT (suprapubic approach); Procedure: Li-SWT (perineal approach); Procedure: Li-SWT (combined approach)
- Sham treatment (Sham Comparator): Patients will be treated by 8 sessions of sham treatment with one week interval, applied through suprapubic and perineal approaches.
  Interventions: Procedure: Sham treatment
- antimuscarinics (Active Comparator): Patients will be treated by solifenacin 10 mg once daily for 6 months.
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Procedure: Li-SWT (suprapubic approach) — The patient will be asked to lie in flat dorsal position. A commercially used gel for sonography will be applied to the suprapubic region. The applicator will be placed on suprapubic region with two fingers apart from the symphysis pubis tilting to 45°. Shock waves will be directed to 3 different sites; the midline (over the bladder dome) and 3 cm right and left to the midline (over bilateral bladder walls). The patient will receive 3000 shocks (1000 shocks per site) with energy flux density of 0.12 mJ/mm² and frequency of 4 Hz.
  Arms: Li-SWT
Procedure: Li-SWT (perineal approach) — The patient will be asked to lie in lithotomy position. A commercially used gel for sonography will be applied to the perineum. The applicator will be placed on perineal region. Shock waves will be directed to 3 different sites: the midline and 2 cm above and below the midline. The patient will receive 3000 shocks (1000 shocks per site) with energy flux density of 0.12 mJ/mm² and frequency of 4 Hz.
  Arms: Li-SWT
Procedure: Li-SWT (combined approach) — The patient will receive 3000 shocks; 1500 shocks through suprapubic approach (500 shocks per site) and another 1500 shocks through perineal approach (500 shocks per site) with energy flux density of 0.12 mJ/mm² and frequency of 4 Hz.
  Arms: Li-SWT
Procedure: Sham treatment — The same technique of Li-SWT will be used but the applicator of the shock wave device will be turned off.
  Arms: Sham treatment
Drug: Solifenacin — The patients will be treated by antimuscarinics (solifenacin) which are considered as the conventional treatment of storage symptoms after prostatectomy.
  Arms: antimuscarinics

SUMMARY:
comparing the outcome of low-intensity shock wave therapy (Li-SWT) versus solifenacin on persistent storage symptoms after transurethral surgery for benign prostatic obstruction (BPO)

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a common cause of lower urinary tract symptoms (LUTS) in aging men including both voiding and storage symptoms. After prostatectomy, 20-30% of the patients still have persistent storage symptoms. The pathophysiology of persistent storage symptoms after surgical relief of benign prostatic obstruction (BPO) remains unclear. It may be due to bladder changes produced by long standing bladder outlet obstruction (BOO) including bladder ischemia and denervation or it may be related to other factors rather than preoperative BOO such as aging, chronic inflammation or a subtle neurological disorder.

After exclusion of urinary tract infection (UTI) and BOO, antimuscarinics are the commonly used medications for post-prostatectomy persistent storage symptoms. However, these medications are associated with side effects which may interfere with the patient compliance.

Low-intensity shock wave therapy (Li-SWT) is a non invasive procedure that has a beneficial effect in promoting revascularization and enhancing tissue regeneration. It has been applied to the penis for erectile dysfunction and to the perineum for chronic pelvic pain syndrome (CPPS) with encouraging results. In a rat model, it has been reported that defocused Li-SWT leads to improvement of bladder innervation and vascularization.

Based on the previously mentioned studies, the investigators hypothesized that Li-SWT can offer benefit in improvement of persistent storage symptoms after surgical relief of BPO. In the present study, the investigators will evaluate the effect of Li-SWT on persistent storage symptoms after transurethral surgery for BPO compared to antimuscarinics in a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients have to fulfill all the following criteria to be included in the study:

  1. Ability to give informed consent and reply to questionnaires.
  2. Average urgency episodes per 24 hrs ≥ 1 and average daytime frequency ≥ 8 during the baseline 3-day voiding diary.
  3. Relief of BOO as proved by non-invasive uroflowmetry, pressure flow study (PFS) or urethrocystoscopy.

Exclusion Criteria:

* Patients who have any of the following will be excluded from the study:

  1. Untreated UTI.
  2. BOO such as bladder neck contracture (BNC), residual obstructing adenoma or urethral stricture.
  3. Neurogenic lower urinary tract dysfunction (LUTD).
  4. Uncontrolled diabetes mellitus.
  5. Depression or any psychogenic disorders.
  6. Prior radiation therapy to the pelvic area.
  7. History of prostate cancer, bladder tumor or intravesical Bacillus Calmette Guerin (BCG) therapy.
  8. Poor coagulopathy.
  9. Severe cardiovascular disease.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients suffering from persistent storage symptoms ≥ 3 months following any transurethral surgery for BPO will be asked to participate in this study.
Enrollment: 132 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
The percent change in overactive bladder symptoms score (OABSS) | approximately 20 months
  The primary endpoint is the percent change from baseline in the total score of OABSS (total score = 15) at 3-month follow up.
Percent of responders | approximately 20 months
  The percent of responders at 3-month follow up. Three points reduction in the total score of OABSS is determined as the minimal threshold for a meaningful change. Responders are defined as patients who achieved reduction in the total score of OABSS ≥ 3 at 3-month follow up, and those patients will continue on the same treatment modality.
The numerical change in overactive bladder symptoms score (OABSS) | approximately 2 years.
  The numerical change from baseline in the total score and sub-scores of OABSS at 3 and 6-month follow up will be reported.
3-day voiding diary | approximately 2 years.
  Change in daytime frequency (times/24hrs), urgency (times/24hrs), urge incontinence (times/24hrs), nocturia (times/24hrs) and average voided volume/micturition (ml) from baseline will be compared at 3 and 6-month follow up.
Incidence of adverse events associated with treatment | approximately 18 months
  Incidence of adverse events associated with Li-SWT or solifenacin (n%) should be reported.

SECONDARY OUTCOMES:
International index of prostate symptom score (IPSS) | approximately 2 years.
  Change in IPSS at 0, 3 and 6 months will be compared.
Post voiding residual urine (PVR) | approximately 2 years.
  Change in PVR (ml) at 0, 3 and 6 months will be compared.
Maximum flow rate (Qmax) | approximately 2 years.
  Change in Qmax (ml/s) at 0, 3 and 6 months will be compared.
International index of erectile function-15 ( IIEF-15) | approximately 2 years.
  Change in IIEF-15) at 0, 3 and 6 months will be compared.
Cystometric bladder capacity | approximately 2 years.
  Change in bladder volume (ml) at first sensation of filling and maximum cystometric capacity (ml) at 0 and 6 months will be analysed.
Detrusor overactivity | approximately 2 years.
  Change in detrusor stability and maximum amplitude (cmH2O) of detrusor overactivity during cystometry at 0 and 6 months will be analysed.
Detrusor contractility | approximately 2 years.
  Change in maximum detrusor pressure (cmH2O) and BCI during voiding at 0 and 6 months will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Hegazy, Principal Investigator — Urology and nephrology center, Mansoura, Egypt; Mohamed Gaballah, Study Director — Urology and nephrology center, Mansoura, Egypt; Khaled Sheir, Study Director — Urology and nephrology center, Mansoura, Egypt; Ahmed Elshal, Study Director — Urology and nephrology center, Mansoura, Egypt
Locations (1):
- Urology and Nephrology center, Al Mansurah, Egypt